CLINICAL TRIAL: NCT03569371
Title: A Phase 2, Open-Label, Single-Arm Study of the Safety of INCB054707 in Participants With Hidradenitis Suppurativa
Brief Title: A Study of the Safety of INCB054707 in Participants With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54707-202
Record Dates: First submitted 2018-05-24; First posted 2018-06-26 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa (HS); Janus kinase (JAK); Janus kinase 1 (JAK1) inhibitor
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB054707 (Experimental)
  Interventions: Drug: INCB054707

INTERVENTIONS:
Drug: INCB054707 — INCB054707 administered once daily orally with water without regard to food for 8 weeks.
  Other Names: Povorcitinib

SUMMARY:
The purpose of this study is to assess the safety of INCB054707 in men and women with moderate to severe hidradenitis suppurativa (HS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS (confirmed by a dermatologist) with a disease duration of at least 6 months before screening.
* Stable course of HS for at least 90 days before screening, as determined by the investigator.
* HS lesions present in at least 2 distinct anatomic areas, 1 of which must be Hurley Stage II or III at screening and baseline.
* Total AN count of at least 3 at screening and baseline.
* Male participants must agree to use contraception per protocol-defined criteria.

Exclusion Criteria:

* Women of childbearing potential or who are currently pregnant or lactating.
* Presence of > 20 draining fistulas at screening and baseline.
* Participants with concurrent conditions or history of other diseases as follows:

  * Any clinically significant medical condition other than HS, as determined by the investigator, that is not adequately controlled with appropriate treatment.
  * Any other active skin disease or condition (eg, bacterial, fungal, or viral infection) that may interfere with the course, severity, or assessments of HS.
  * Active systemic viral infection or any active viral infection that, based on the investigator's clinical assessment, make the participant an unsuitable candidate for the study.
  * Current herpes zoster infection, a history of recurrent herpes zoster, a history of disseminated herpes simplex, or a history of herpes zoster.
  * History of malignancy, including lymphoma and leukemia within 5 years before baseline, other than a successfully treated nonmetastatic cutaneous squamous cell carcinoma, basal cell carcinoma, or localized carcinoma in situ of the cervix.
  * Albinism.
* Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF), defined as ≥ 450 msec.
* Positive test result for tuberculosis (TB) from the QuantiFERON-TB Gold test, or equivalent, at screening (or, if 2 indeterminate tests or not available, then as evaluated by a purified protein derivative test with a result of < 5 mm of induration within 3 months of screening) or a history of active TB.
* Positive serology test results for HIV, HBsAg, hepatitis B virus (HBV) core antibody, or HCV (HCV antibody with positive HCV-RNA) at screening.
* Decreased blood cell counts at screening as per protocol-defined parameters.
* Severely impaired liver function (Child-Pugh Class C) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels ≥ 1.5 × upper limit of normal (ULN).
* Impaired renal function with serum creatinine > 1.5 mg/dL.
* Use of prohibited medications per protocol-defined criteria.
* Known or suspected allergy to INCB054707 or any component of the study drug.
* Known history of clinically significant drug or alcohol abuse in the last year prior to baseline.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (4):
- United States (4):
  - Investigative Site, Los Angeles, California
  - Investigative Site, Tampa, Florida
  - Investigative Site, New York, New York
  - Investigative Site, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alavi A, Hamzavi I, Brown K, Santos LL, Zhu Z, Liu H, Howell MD, Kirby JS. Janus kinase 1 inhibitor INCB054707 for patients with moderate-to-severe hidradenitis suppurativa: results from two phase II studies. Br J Dermatol. 2022 May;186(5):803-813. doi: 10.1111/bjd.20969. Epub 2022 Mar 6. PMID 34978076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 different sites in US.
Pre-assignment Details: A total of 10 participants were assigned to treatment with INCB054707.
Groups:
- INCB054707: Participants were treated with 15 mg QD of INCB054707 orally.
Period: Overall Study
Arm/Group | INCB054707
Started | 10
Completed | 7
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Number] | 40.7 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 6
  Black/African American | 3
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Time Frame: Up to approximately 12 weeks.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Number; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants | 7

2. Secondary Outcome: Apparent Oral Clearance of INCB054707(CL/F)
Description: To evaluate the systemic exposure to INCB054707.
Time Frame: Postdose Day1, week 2 and 6
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | INCB054707
Number analyzed (Participants) | 10
L/hr | 5.07 (24.3)

3. Secondary Outcome: Apparent Oral Volume of Distribution of INCB054707(Vc/F)
Description: To evaluate the systemic exposure to INCB054707.
Time Frame: Postdose Day1, week 2 and 6.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | INCB054707
Number analyzed (Participants) | 10
L | 227 (39.9)

4. Secondary Outcome: Absorption Constant of INCB054707 (Ka)
Description: Other population pharmacokinetic (PK) model parameter that the PK model may include to evaluate the systemic exposure to INCB054707.
Time Frame: Postdose Day1, week 2 and 6.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | INCB054707
Number analyzed (Participants) | 10
1/hr | 0.257 (15.2)

5. Secondary Outcome: Apparent Inter-compartmental Clearance(Q/F)
Description: Other population PK model parameter that the PK model may include to evaluate the systemic exposure to INCB054707.
Time Frame: Postdose Day1, week 2 and 6.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | INCB054707
Number analyzed (Participants) | 10
L/hr | 16.2 (13.4)

6. Secondary Outcome: Proportion of Participants With a Hidradenitis Suppurativa Clinical Response (HiSCR) at Each Visit
Description: An HiSCR is defined as at least 50% reduction in abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline at each visit.
Time Frame: Weeks 1,2,4,6,8 and FollowUp
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Week 1: number analyzed (Participants) | 9
  Week 1 | 1
  Week 2: number analyzed (Participants) | 9
  Week 2 | 3
  Week 4: number analyzed (Participants) | 9
  Week 4 | 3
  Week 6: number analyzed (Participants) | 7
  Week 6 | 2
  Week 8: number analyzed (Participants) | 7
  Week 8 | 3
  Follow Up: number analyzed (Participants) | 7
  Follow Up | 4

7. Secondary Outcome: Proportion of Participants Achieving an AN Count of 0 to 2 at Each Visit
Description: The number and proportion of participants who achieved an Abscess and Inflammatory nodule count of 0 to 2 progressively.
Time Frame: Weeks 1,2,4,6,8 and FollowUp
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Baseline | 0
  Week 1: number analyzed (Participants) | 9
  Week 1 | 2
  Week 2: number analyzed (Participants) | 9
  Week 2 | 4
  Week 4: number analyzed (Participants) | 9
  Week 4 | 4
  Week 6: number analyzed (Participants) | 7
  Week 6 | 2
  Week 8: number analyzed (Participants) | 7
  Week 8 | 3
  Follow Up: number analyzed (Participants) | 7
  Follow Up | 4

8. Secondary Outcome: Mean Change From Baseline in the HS Pain Numeric Rating Scale (NRS) Scores at Each Visit
Description: The HS Pain NRS will be completed in a daily diary by participants from screening through EOS. An 11-point scale will be used to assess the worst skin pain due to HS based on a recall period of the last 24 hours. Ratings for the 2 items range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine)
Time Frame: Weeks 1,2,4,6,8 and FollowUp
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Units on a Scale
  Week 1 | -1.5 (1.9)
  Week 2: number analyzed (Participants) | 9
  Week 2 | -3.2 (2.9)
  Week 4: number analyzed (Participants) | 9
  Week 4 | -2.6 (2.9)
  Week 6: number analyzed (Participants) | 7
  Week 6 | -3.2 (3.2)
  Week 8: number analyzed (Participants) | 7
  Week 8 | -2.0 (1.8)
  Follow Up: number analyzed (Participants) | 6
  Follow Up | -1.8 (1.6)

9. Secondary Outcome: Mean Change From Baseline in the Modified Sartorius Scale Score
Description: The Sartorius Scale is used to quantify the severity of HS. Points are awarded for 12 body areas (left and right axillae, left and right sub/inframammary areas, intermammary area, left and right buttocks, left and right inguino-crural folds, perianal area, perineal area, and other). For each area, points are awarded for nodules (2 points for each); abscesses (4 points); fistulas (4 points); scars (1 point); longest distance between two lesions (2-6 points, 0 if no lesions); and if lesions are separated buy normal skin (yes-0 point; no-6 points). The total Sartorius Scale score is the sum of the 12 regional scores. Scale scores range from 0 to infinite, with larger scores representing higher severity of HS.
Time Frame: Week 8.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Units on a Scale | -13.6 (21.3)

10. Secondary Outcome: Mean Change From Baseline in the Number of Draining Fistulas Count at Each Visit
Description: Draining fistulas are fistulas that drain serous or purulent fluid, either spontaneously or by gentle palpation.
Time Frame: Up to approximately 12 weeks.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Mean (Standard Deviation); unit: Number of Fistulas
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Number of Fistulas
  Week 1: number analyzed (Participants) | 9
  Week 1 | -0.1 (0.6)
  Week 2: number analyzed (Participants) | 9
  Week 2 | 0.2 (0.4)
  Week 4: number analyzed (Participants) | 9
  Week 4 | 0.6 (1.7)
  Week 6: number analyzed (Participants) | 7
  Week 6 | 1.9 (2.9)
  Week 8: number analyzed (Participants) | 7
  Week 8 | 0.1 (1.1)
  Follow Up: number analyzed (Participants) | 7
  Follow Up | 0.7 (2.4)

11. Secondary Outcome: Proportion of Participants at Each Category of Hurley Stage
Description: The Hurley classification is a static score and was originally designed for selection of the appropriate treatment modality in a certain body region. The assessor determines the Hurley stage in each affected anatomical region. If more than 1 stage is present in the same region, the worst stage in that region is documented. The participant will be assigned an overall Hurley stage classification corresponding to the stage of the worst involved anatomical region. The definition of each Hurley stage is as follows:
  Stage I : Abscess formation, single or multiple, without sinus tracts and cicatrization (scarring).
  Stage II : One or more widely separated recurrent abscesses with tract formation and cicatrization (scarring).
  Stage III : Multiple interconnected tracts and abscesses across the entire area, with diffuse or near diffuse involvement.
Time Frame: Baseline and Week 8.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Baseline: Stage I | 0
  Baseline: Stage II | 7
  Baseline: Stage III | 3
  Baseline: No HS | 0
  Week 8: number analyzed (Participants) | 7
  Week 8: Stage I | 0
  Week 8: Stage II | 5
  Week 8: Stage III | 1
  Week 8: No HS | 1

12. Secondary Outcome: Proportion of Participants With Change From Baseline to Week 8 in Hurley Stage
Description: as for outcome 11
Time Frame: Week 8.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Baseline: No HS | 0
  Baseline: Stage I | 0
  Baseline: Stage II | 7
  Baseline: Stage III | 3
  Week 8: number analyzed (Participants) | 7
  Week 8: No HS | 1
  Week 8: Stage I | 0
  Week 8: Stage II | 5
  Week 8: Stage III | 1

13. Secondary Outcome: Proportions of Participants in Each HS Patient Global Impression of Change (PGIC) Category
Description: The HS-PGIC consists of 1 self-administered item that assesses change in the severity of skin in the HS area. The participant will answer the following: Since your last visit, your HS is: (1) very much improved, (2) much improved, (3) minimally improved, (4) no change, (5) minimally worse, (6) much worse, or (7) very much worse.
Time Frame: Up to approximately 12 weeks.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Week 1: 1 | 0
  Week 1: 2 | 0
  Week 1: 3 | 3
  Week 1: 4 | 5
  Week 1: 5 | 2
  Week 1: 6 | 0
  Week 1: 7 | 0
  Week 2: number analyzed (Participants) | 9
  Week 2: 1 | 0
  Week 2: 2 | 1
  Week 2: 3 | 5
  Week 2: 4 | 2
  Week 2: 5 | 1
  Week 2: 6 | 0
  Week 2: 7 | 0
  Week 4: number analyzed (Participants) | 9
  Week 4: 1 | 1
  Week 4: 2 | 1
  Week 4: 3 | 0
  Week 4: 4 | 4
  Week 4: 5 | 3
  Week 4: 6 | 0
  Week 4: 7 | 0
  Week 6: number analyzed (Participants) | 7
  Week 6: 1 | 1
  Week 6: 2 | 1
  Week 6: 3 | 2
  Week 6: 4 | 2
  Week 6: 5 | 1
  Week 6: 6 | 0
  Week 6: 7 | 0
  Week 8: number analyzed (Participants) | 7
  Week 8: 1 | 0
  Week 8: 2 | 1
  Week 8: 3 | 2
  Week 8: 4 | 3
  Week 8: 5 | 1
  Week 8: 6 | 0
  Week 8: 7 | 0
  Follow Up: number analyzed (Participants) | 6
  Follow Up: 1 | 0
  Follow Up: 2 | 1
  Follow Up: 3 | 2
  Follow Up: 4 | 3
  Follow Up: 5 | 0
  Follow Up: 6 | 0
  Follow Up: 7 | 0

14. Secondary Outcome: Proportion of Participants Requiring Rescue Lesional Treatment
Description: Rescue lesional treatment is defined as immediate intervention in the event of an acutely painful lesion.
Time Frame: Up to approximately 12 weeks.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Week 1: Intervention Required -Yes | 1
  Week 1: Intervention Required -No | 9
  Week 2: number analyzed (Participants) | 9
  Week 2: Intervention Required -Yes | 0
  Week 2: Intervention Required -No | 9
  Week 4: number analyzed (Participants) | 9
  Week 4: Intervention Required -Yes | 0
  Week 4: Intervention Required -No | 9
  Week 6: number analyzed (Participants) | 7
  Week 6: Intervention Required -Yes | 0
  Week 6: Intervention Required -No | 7
  Week 8: number analyzed (Participants) | 7
  Week 8: Intervention Required -Yes | 1
  Week 8: Intervention Required -No | 6
  Follow Up: number analyzed (Participants) | 7
  Follow Up: Intervention Required -Yes | 0
  Follow Up: Intervention Required -No | 7

15. Secondary Outcome: Number of Interventions With Rescue Lesional Treatment
Description: Rescue lesional treatment is defined as immediate intervention in the event of an acutely painful lesion.
Time Frame: Up to approximately 12 weeks.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Mean (Standard Deviation); unit: Interventions
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Interventions
  Week 1 | 0.1 (0.32)
  Week 2: number analyzed (Participants) | 9
  Week 2 | 0 (0.00)
  Week 4: number analyzed (Participants) | 9
  Week 4 | 0 (0.00)
  Week 6: number analyzed (Participants) | 7
  Week 6 | 0 (0.00)
  Week 8: number analyzed (Participants) | 7
  Week 8 | 0.1 (0.38)
  Follow Up: number analyzed (Participants) | 7
  Follow Up | 0 (0.00)

16. Secondary Outcome: Proportion of Participants at Each Scoring Category of the Dermatology Life Quality Index (DLQI) at Each Visit
Description: The DLQI is a questionnaire used to assess the symptoms and the impact of skin problems on quality of life. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The meaning of DLQI scores can be categorized as follows: 0-1 = No effect at all on patient's life 2-5 = Small effect on patient's life 6-10 = Moderate effect on patient's life 11-20 = Very large effect on patient's life 21-30 = Extremely large effect on patient's life
Time Frame: Up to approximately 12 weeks.
Population: The Full Analysis Set population include all subjects enrolled in the study who received at least 1 dose of INCB054707
Measure: Count of Participants; unit: Participants
Arm/Group | INCB054707
Number analyzed (Participants) | 10
Participants
  Baseline: 0-1 | 0
  Baseline: 2-5 | 1
  Baseline: 6-10 | 3
  Baseline: 11-20 | 2
  Baseline: 21-30 | 4
  Week 1: 0-1 | 0
  Week 1: 2-5 | 2
  Week 1: 6-10 | 2
  Week 1: 11-20 | 3
  Week 1: 21-30 | 3
  Week 2: number analyzed (Participants) | 9
  Week 2: 0-1 | 0
  Week 2: 2-5 | 5
  Week 2: 6-10 | 1
  Week 2: 11-20 | 1
  Week 2: 21-30 | 2
  Week 4: number analyzed (Participants) | 9
  Week 4: 0-1 | 2
  Week 4: 2-5 | 1
  Week 4: 6-10 | 2
  Week 4: 11-20 | 3
  Week 4: 21-30 | 1
  Week 6: number analyzed (Participants) | 7
  Week 6: 0-1 | 1
  Week 6: 2-5 | 1
  Week 6: 6-10 | 2
  Week 6: 11-20 | 1
  Week 6: 21-30 | 2
  Week 8: number analyzed (Participants) | 7
  Week 8: 0-1 | 0
  Week 8: 2-5 | 3
  Week 8: 6-10 | 1
  Week 8: 11-20 | 1
  Week 8: 21-30 | 2
  Follow Up: number analyzed (Participants) | 7
  Follow Up: 0-1 | 0
  Follow Up: 2-5 | 3
  Follow Up: 6-10 | 0
  Follow Up: 11-20 | 2
  Follow Up: 21-30 | 2

ADVERSE EVENTS:
Time Frame: Up to approximately 12 weeks
Arm/Group | INCB054707
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INCB054707 (N=10)
Nausea (Gastrointestinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03569371/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT03569371/SAP_001.pdf